CLINICAL TRIAL: NCT04650425
Title: Causal Evidence for Task Regulation by Anterior Cingulate Cortex
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Ghent (Other)
Collaborators: Neurology (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-08764
Record Dates: First submitted 2020-11-12; First posted 2020-12-02 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: Anterior Cingulate Cortex
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Each participant will undergo one or two sessions, consisting of cognitive tasks, video-EEG recording and administering of questionnaires.
  Interventions: Behavioral: Cognitive tasks

INTERVENTIONS:
Behavioral: Cognitive tasks — Patients will perform the coffee-tea task and the virtual T-maze task, both in the acute and chronic phase after stroke.

SUMMARY:
The exact function of the anterior cingulate cortex (ACC) is one of the largest riddles in cognitive neuroscience and a major challenge in mental health research. ACC dysfunction contributes to a broad spectrum of neurological and psychiatric disorders, such as depression, ADHD, Parkinson's disease, OCD and many others, but nobody knows what it actually does. Recently a new theory has been developed about ACC function; the HRL-ACC (Hierarchical Reinforcement Learning Theory of ACC). This theory proposes that the ACC selects and motivates high-level tasks based on the principles of hierarchical reinforcement learning. The ACC associates values with tasks (these values are based on the reward positivity produced by the midbrain dopamine system), selects the correct tasks and applies control over other neural networks (such as the dorsolateral prefrontal cortex and basal ganglia), which execute the tasks. The goal of this study is to investigate the consequences of ACC damage (and other areas of the frontal lobe) on task regulation within a group of patients who have suffered a stroke in the frontal lobe. Furthermore, the correlation between ACC damage and mood disorders such as depression and apathy is going to be investigated.

DETAILED DESCRIPTION:
This is a monocentric prospective interventional clinical trial that will include patients with a stroke in the frontal lobe. Depending on the recruitment manner, participants will undergo one or two sessions of cognitive experiments. The patients will be recruited in two ways, through the Stroke unit and through the outpatient clinic:

1. If a patient with an acute stroke in the frontal lobe is admitted to the Stroke unit and is eligible for this study, the patient will be asked if he is willing to participate. After giving informed consent, the first session will take place once the patient has been transferred to a regular neurological ward. After discharge, a second session will take place 6 to 12 months later at the outpatient clinic, preferably combined with a consultation (as part of the standard of care of stroke patients).
2. Patients who have had a stroke are followed at the outpatient clinic. Patients who are eligible for this study, will be contacted by the treating stroke supervisor during their consultation (either Prof. Veerle De Herdt or Dr. Dimitri Hemelsoet). If they are willing to participate, the first session will take place either right after the consultation at the outpatient clinic, or - if the patient is not available at that time - a new appointment will be made.

One experimental session consists of the following steps:

* Clinical neurological examination with determining of NIHSS score.
* First cognitive task: the coffee-tea task. During this task, a sequence of 7 images is shown and each image contains three objects. The patient has to choose the right objects to make either coffee or tea. At the end of each sequence they get feedback if they have prepared the beverage correctly or not.
* Short break with positioning of 21 EEG electrodes.
* Second task: the virtual T-maze task with video-EEG recording. During this task, a virtual T-maze is shown and the patient has to choose at each junction whether they go left or right. Depending on which direction they choose, they either get positive or negative feedback. This task is known to elicit the reward positivity. During this task, video-EEG will be recorded and this EEG-data will later on be analysed using ERP analysis.
* If second session, administering of questionnaires: Oxford Cognitive Screen, Becker Depression Inventory, DEX apathy questionnaire.

Furthermore, the investigators are going to use voxel-based lesion symptom mapping to analyze the relationship between tissue damage and behavioural problems and reward positivity amplitude.

It is expected that the coffee-tea task will be more difficult for patients with ACC damage compared to patients with lesions in other areas of the frontal lobe. Also, the amplitude of the ERP signals during the virtual T-maze task will be smaller in patients with ACC damage. Furthermore, the investigators expect to find a connection between ACC damage and mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patients: ischemic stroke or intracranial hemorrhage
* Involvement of the frontal lobe
* Lesion is visible on CT and/or MRI and is concordant with clinical presentation during the time of onset
* Patients have to be able to give informed consent themselves

Exclusion Criteria:

* Patients with a TIA, i.e. no visible lesion on CT and/or MRI or symptoms less than 24 hours
* Patients with decreased alertness or disorders of consciousness, which makes it impossible for these patients to participate in the experiments
* Active alcohol and/or drug abuse/addiction
* Patients diagnosed with dementia or another neurodegenerative disease, or severe cognitive and/or psychiatric disorders that make it impossible for these patients to participate in the study
* Patients with severe aphasia (as defined by NIHSS score)
* A history of stroke in the frontal lobe is NOT an exclusion criteria (except when the patient has been diagnosed with poststroke frontal dysfunction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and type of mistakes made during the coffee-tea task | date of inclusion to date of second session, assessed up to 6 to 12 months
  Analysed and compared within sub-groups (classified by using Voxel-based Lesion Symptom Mapping)
Amplitude of reward positivity Event-Related Potential signals | date of inclusion to date of second session, assessed up to 6 to 12 months
  Relationship between reward positivity amplitude and brain damage, investigated by using Voxel-based Lesion Symptom Mapping.
Neurofunctional status | 6 to 12 months after stroke
  Neurofunctional status as defined by the Oxford Cognitive Score, a scale ranging from 0 to 138 (the higher the score, the better the neurofunctional status)
Presence of depression | 6 to 12 months after stroke
  Presence and severity of depression, evaluated by using the Becker Depression Inventory, a scale that scores from 0 to 63 (the higher the score, the more severe the depression).
Presence of apathy | 6 to 12 months after stroke
  Presence and severity of apathy, evaluated by using the DEX (Dysexecutive) Questionnaire, a scale that scores from 0 to 80 and that is filled in both by the patient and the independent caretaker (e.g. family, friend). The higher the score, the more severe the apathy and dysexecutive problems.

SECONDARY OUTCOMES:
Performance of coffee-tea task in subgroup with ACC lesions | date of inclusion to date of second session, assessed up to 6 to 12 months
  Comparing the results of the coffee-tea task performed by the ACC-subgroup to the results of the other subgroups, by using Voxel-based Lesion Symptom Mapping, and therefore assessing the crucial role of ACC on task regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle De Herdt, Principal Investigator — University Hospital Ghent, Department of Neurology
Locations (1):
- University Hospital, department of neurology, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided